CLINICAL TRIAL: NCT00664794
Title: Arthroscopic Rotator Cuff Repair With and Without Arthroscopic Acromioplasty in the Treatment of Full Thickness Rotator Cuff Tears
Brief Title: Rotator Cuff Repair With Arthroscopic Acromioplasty (Shaving the Acromion Bone) Versus Repair Without Acromioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005883-01H
Record Dates: First submitted 2008-01-21; First posted 2008-04-23 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without acromioplasty (Active Comparator)
  Interventions: Procedure: without acromioplasty
- with acromioplasty (Active Comparator)
  Interventions: Procedure: with acromioplasty

INTERVENTIONS:
Procedure: without acromioplasty — This group will not have their acromion shaved - instead they will receive a repair of their rotator cuff with the scope using sutures or suture anchors.
  Arms: without acromioplasty
Procedure: with acromioplasty — This group will have Their rotator cuff repaired with sutures or suture anchors and additionally will have the tip of their acromion bone shaved slightly.
  Arms: with acromioplasty

SUMMARY:
Surgical repair of full-thickness tears of the rotator cuff is a controversial issue, with several procedures currently being used to treat the tear. The two most common treatments at this point in time are arthroscopic cuff repair with and without acromioplasty. However, an arthroscopic cuff repair without acromioplasty may offer the same degree of improvement as one that includes acromioplasty, but without threatening the shoulder stability that is provided by the acromion and coracoacromial ligament. This prospective study examines the hypothesis that appropriate shoulder function can be restored through execution of the traditional arthroscopic cuff repair without acromioplasty.

DETAILED DESCRIPTION:
The rotator cuff is a musculotendinous amalgamation of four muscles that arise from the scapula and insert on the proximal humerus. The tendons of the supraspinatus, infraspinatus, subscapularis, and teres minor form a continuous cuff around the humeral head and allow for a variety of movements in rotation of the humeral head. Tears of one or more of these tendons that comprise the rotator cuff are one of the many causes of pain and disability in the shoulder12. Treatment of these tears has included both operative and non-operative approaches. The non-operative approaches have generally included modification of activities, administration of analgesic or anti-inflammatory medication, and a progressive physiotherapy program aimed at regaining a full range of motion about the shoulder and full strength in the rotator cuff. The results stemming from this treatment have for the most part been disappointing 13.

Codman16 was the first to describe an open surgical technique for rotator cuff repair and Neer17 later refined the existing surgical technique in addition to being the first to apply acromioplasty to repair of tears of the rotator cuff. Since that time, operative repair of full-thickness tears of the rotator cuff has gradually shifted from open repair to arthroscopic repair with some combined open/arthroscopic (mini-open) procedures being performed. The mini-open procedure involves arthroscopic evaluation of the glenohumeral joint and arthroscopic acromioplasty coupled with open repair of the cuff tear15. As surgeons gained experience with the mini-open repair, they began to familiarize themselves with the arthroscopic appearance of rotator cuff tears and improved their ability to arthroscopically measure the tear and assess its repairability4. These advances combined with improvements in arthroscopic instruments and suturing techniques have allowed the elimination of the open portion of the mini-open repair and the emergence of a completely arthroscopic procedure. Exclusive arthroscopic repair of rotator cuff tears provides the advantages of deltoid preservation, less soft tissue dissection, shortened hospital stay, and accelerated rehabilitation. It also allows for visualization of the glenohumeral joint, which can be advantageous since several authors have reported a 60-75 % incidence of coinciding glenohumeral pathologies with cuff tears5,6.

There exists some controversy in the current trend in repair of full-thickness tears of the rotator cuff. The two most common treatments at this point in time are arthroscopic cuff repair with and without acromioplasty. The purpose of acromioplasty is to create adequate space for the rotator cuff tendons. Arthroscopic acromioplasty involves removal of the subacromial bursa, resection of the coracoacromial ligament and anteroinferior portion of the acromion, and resection of any osteophytes from the acromioclavicular joint that are thought to be contributing to impingement. However, acromioplasty without cuff repair has been reported to have both good9,10 and poor11,14 results, showing that the technique may be suspect in repair of full-thickness tears alone.

Budoff and his colleagues have suggested that since the coracoacromial ligament stabilizes the rotator cuff to prevent uncontrolled migration of the humeral head, resection of the coracoacromial ligament during arthroscopic acromioplasty may cause additional long-term migration of the humeral head7. Likewise, Nirschl has suggested that the coracoacromial ligament be resected only in those cases with a specific pathological indication relating to the coracoacromial ligament8. He also states that, "there is no evidence to support the belief that failure to resect the coracoacromial ligament compromises the success of rotator cuff surgery."

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older
* Diagnosis of full-thickness rotator cuff tear
* Ability to understand and adhere to rehab protocols and testing procedure
* Persistent pain and functional disability for at least 6 months and failure of 6 months of conservative treatment

Exclusion Criteria Preoperative

* Evidence of significant osteoarthritis or cartilage damage in the shoulder
* Evidence of glenohumeral instability including Bankart lesions and labral tears of any type
* Previous surgeries of the shoulder
* Evidence of major joint trauma, infection, or necrosis in the shoulder
* Patients with partial-thickness tears of the rotator cuff
* Patients unable to provide informed consent due to language barrier or mental status
* Patients with a major medical condition that would affect quality of life and influence the results of the study
* Patients with worker compensation claims
* Patients unwilling to be followed for the duration of the study.

Patient is automatically ineligible for study if 1 or more exclusion criteria is present.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Determine clinical impact by comparing the intervention and control sites for: | Feb 2008
Patient satisfaction | end of study

SECONDARY OUTCOMES:
Determine sustainability of the impact; | end of study
Accuracy | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Study Chair — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - Pan Am Clinic Foundation, Winnipeg, Manitoba
  - The Ottawa Hospital, Ottawa, Ontario

REFERENCES:
- [Result] MacDonald P, McRae S, Leiter J, Mascarenhas R, Lapner P. Arthroscopic rotator cuff repair with and without acromioplasty in the treatment of full-thickness rotator cuff tears: a multicenter, randomized controlled trial. J Bone Joint Surg Am. 2011 Nov 2;93(21):1953-60. doi: 10.2106/JBJS.K.00488. PMID 22048089